CLINICAL TRIAL: NCT02770742
Title: Patient Satisfaction With Sedated vs. Unsedated Colonoscopy - Which Factors Affect Satisfaction and Pain in Routine Care?
Brief Title: Patient Satisfaction With Sedated vs. Unsedated Colonoscopy
Status: Completed | Type: Observational
Sponsor: Helios Research Center (Other)
Responsible Party: Principal Investigator, Alexander Eckardt, MD, PD Dr. med. Alexander Eckardt, Helios Research Center
Other Study IDs: HRC[058465]
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Satisfaction
Keywords: patient satisfaction; unsedated colonoscopy; intestinal diseases
MeSH Terms: conditions — Personal Satisfaction; Patient Satisfaction; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients for outpatient colonoscopy: The cohort consists of subsequent patients who present for routine colonoscopy. There is no active Intervention. However, groups who choose to perform colonoscopy with or without sedation will be compared.

SUMMARY:
This is a prospective, observational study to evaluate patient satisfaction with colonoscopy, depending on whether sedation is used during the procedure or not. Patients will receive questionnaires before the procedure to assess the potential influence of patient criteria and after the procedure to assess satisfaction-scores and pain-scores. A validated satisfaction score (Schoen et al.) will be used for the primary outcome. As secondary parameters, pain- and sedation-scores will be assessed by the validated NAPCOMS score, as well as procedural quality indicators. The study will assess, whether adequate selection in regards to risk factors for sedated or unsedated colonoscopy, leads to similar satisfaction-scores within both groups.

DETAILED DESCRIPTION:
This is a prospective, observational study of consecutive patients presenting for outpatient colonoscopy in a tertiary care hospital with a large ambulatory care section (DKD Helios Klinik Wiesbaden). The primary endpoint of the study is the comparison of a validated patient satisfaction score in patients undergoing colonoscopy with or without sedation. The aim is to assess whether patients, who are deemed appropriate for an unsedated procedure by predefined risk factors and who wish to avoid sedation, will have similar satisfaction scores, as those who undergo sedation. As secondary aims, pain scores (validated NAPCOMS score) and markers of procedural quality (such as completion rates or withdrawal times) will be assessed.

Considering a 2-point difference in the 15-point satisfaction score as clinically relevant and suspecting a 7:3 distribution of procedures with and without sedation, respectively, 1070 patients must be included (at least 749 sedated and 321 unsedated) in order to reach a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting for colonoscopy
* Age >18 years

Exclusion Criteria:

* Patients not giving written consent
* Colonic stenosis or suspected Stenosis
* Active inflammatory bowel disease
* Previous partial resection of the colon
* Polyposis syndromes
* Inability to speak German or fill out a questionnaire in German language
* Vulnerable patients (prisoners, pregnant women, patients with mental retardation, which would affect filling out a questionnaire or answering questions)
* American Society of Anesthesiology (ASA) grade > III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, presenting for outpatient colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2016-10; Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction-score (Schoen et al.) | within 1-2 weeks after the procedure
  The satisfaction score is based on the following three statements: (a) "I was very satisfied with the care I received"; (b) "I would strongly recommend this procedure to friends who qualify for it"; (c) "I would be willing to repeat the exam in the future if necessary." Each statement is coded on a 5-point ordinate scale that includes the following choices: strongly agree, agree, not sure, disagree and strongly disagree. The average of the scores for the three statements will be used as the satisfaction score.

SECONDARY OUTCOMES:
NAPCOMS score | within the procedure and modified 1-2 weeks after the procedure.
  The NAPCOMS was designed to be completed by the endoscopy nurse assisting during the procedure. It is a composite measure that includes 3 domains: pain, sedation, and a global subjective assessment of tolerability.
  The pain domain is defined by using the dimensions of intensity, frequency, and duration, which are each rated with a score from 0 (no occurrence) to 3 (severe, frequent, or prolonged). Sedation is rated according to level of consciousness ranging from 0 (wide awake) to 3 (unconscious), whereas the global tolerability score is rated from 0 (very well tolerated) to 3 (poorly tolerated). The Overall NAPCOMS was defined as the sum of the severity, frequency, and duration of pain domains. Level of sedation and overall global tolerability ratings are assessed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Eckardt, MD, Principal Investigator — DKD Helios Klinik Wiesbaden, Germany
Locations (1):
- DKD Helios Klinik Wiesbaden, Wiesbaden, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckardt VF, Kanzler G, Schmitt T, Eckardt AJ, Bernhard G. Complications and adverse effects of colonoscopy with selective sedation. Gastrointest Endosc. 1999 May;49(5):560-5. doi: 10.1016/s0016-5107(99)70382-2. PMID 10228252
- [Background] Petrini JL, Egan JV, Hahn WV. Unsedated colonoscopy: patient characteristics and satisfaction in a community-based endoscopy unit. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):567-72. doi: 10.1016/j.gie.2008.10.027. PMID 19231501
- [Background] Eckardt AJ, Swales C, Bhattacharya K, Wassef WY, Phelan NP, Zubair S, Martins N, Patel S, Moquin B, Anwar N, Leung K, Levey JM. Open access colonoscopy in the training setting: which factors affect patient satisfaction and pain? Endoscopy. 2008 Feb;40(2):98-105. doi: 10.1055/s-2007-995469. PMID 18253904
- [Background] Cockburn J, Hill D, Irwig L, De Luise T, Turnbull D, Schofield P. Development and validation of an instrument to measure satisfaction of participants at breast screening programmes. Eur J Cancer. 1991;27(7):827-31. doi: 10.1016/0277-5379(91)90126-x. PMID 1834111
- [Background] Schoen RE, Weissfeld JL, Baum A. Development of a simple instrument to measure patient satisfaction with flexible sigmoidoscopy. Gastroenterology 1995; 108: A34